CLINICAL TRIAL: NCT03392064
Title: A Phase 1 Study Evaluating the Safety, Tolerability and Efficacy of AMG 119 in Subjects With Relapsed/Refractory Small Cell Lung Cancer
Brief Title: A Phase 1 Study Evaluating the Safety, Tolerability and Efficacy of AMG 119 in Subjects With RR SCLC
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Study on enrollment hold, may potentially resume. No active subjects on trial.
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20170124
Record Dates: First submitted 2018-01-02; First posted 2018-01-05 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Small Cell Lung Cancer
Keywords: AMG 119; CART; DLL3
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AMG 119 Treatment (Experimental): AMG 119 administered as a one-time intravenous infusion at different cell dose levels
  Interventions: Biological: AMG 119

INTERVENTIONS:
Biological: AMG 119 — Investigational, adoptive cellular immunotherapy for the treatment of small cell lung cancer

SUMMARY:
A study to evaluate the safety and tolerability of AMG 119 in adult subjects with Relapsed/Refractory Small Cell Lung Cancer (SCLC) and determine the appropriate cell dose.

DETAILED DESCRIPTION:
This is a phase 1, first-in-human study to evaluate the safety and tolerability of AMG 119, an investigational, Chimeric Antigen Receptor T cell therapy targeting delta-like protein 3 (DLL3) in subjects with relapsed/refractory small cell lung cancer who progressed after at least 1 platinum based chemotherapy regimen.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided informed consent prior to initiation of any study-specific activities/procedures;
* Age ≥ 18 years old at the time of signing the informed consent
* Histologically or cytologically confirmed Small Cell Lung Cancer (SCLC) with radiographically documented disease progression or recurrence after at least one platinum-based regimen:
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* At least 2 measurable lesions as defined per modified RECIST 1.1 by CT or MRI performed after the last line of anti-cancer therapy within 28 days of enrollment. Subjects with 1 measurable lesion may be considered upon agreement with Sponsor
* Subjects with treated brain metastases are eligible provided they meet the following criteria:
* - Definitive therapy was completed at least 2 weeks prior to enrollment.
* - No evidence of radiographic CNS progression or CNS disease following definitive therapy and by the time of study screening. Patients manifesting progression in lesions previously treated with stereotactic radiosurgery may still be eligible if pseudoprogression can be demonstrated by appropriate means and after discussion with the medical monitor.
* - Any CNS disease is asymptomatic, any neurologic symptoms due to CNS disease have returned to baseline or are deemed irreversible, the patient is off steroids for at least 7 days (physiologic doses of steroids are permitted), and the patient is off or on stable doses of anti-epileptic drugs for malignant CNS disease for at least 7 days.
* Adequate organ function
* Other inclusion criteria may apply

Exclusion Criteria:

* History of other malignancy within the past 2 years prior to enrollment except: Malignancy (other than in situ) treated with curative intent and with no known active disease present for ≥ 2 years before enrollment and felt to be at low risk for recurrence by the treating physician; Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease; Adequately treated in situ cancer without evidence of disease; Prostatic intraepithelial neoplasia without evidence of prostate cancer; Adequately treated urothelial papillary noninvasive carcinoma.
* History of organ transplant.
* Major surgery within 28 days of enrollment.
* Myocardial infarction and/or symptomatic congestive heart failure (New York Heart Association > class II) within 12 months of enrollment.
* History of arterial thrombosis (eg, stroke or transient ischemic attack) within 12 months of enrollment.
* Untreated or symptomatic brain metastases and leptomeningeal disease
* Presence of fungal, bacterial, viral, or other infection requiring IV antimicrobials for management within 7 days of enrollment. Note: Simple UTI and uncomplicated bacterial pharyngitis are permitted if responding to active treatment and after consultation with sponsor.
* Known sensitivity and immediate hypersensitivity to any components of AMG 119 or conditioning regimen (cyclophosphamide and fludarabine).
* Evidence of a bleeding diathesis.
* Systemic corticosteroid therapy within 7 days before enrollment. Note: Topical and inhaled corticosteroids in standard doses and physiologic replacement for subjects with adrenal insufficiency are allowed. ≥ 5 mg/day of prednisone or equivalent doses of other corticosteroids are not allowed.
* Prior anti-cancer therapy as specified below: At least 21 days from enrollment must have elapsed from any prior systemic inhibitory/stimulatory immune checkpoint molecule therapy (eg, ipilimumab, nivolumab, pembrolizumab, atezolizumab, OX40 agonists, 4-1BB agonists, etc). Note: Patients who experienced immune -related pneumonitis, pituitary or thyroid dysfunction, or pancreatitis while on treatment with immune-oncology agents will be excluded; Other anti-cancer therapy (chemotherapy, antibody therapy, molecular targeted therapy, or investigational agent) within 14 days prior to enrollment; Radiation therapy completed within 14 days prior to enrollment; Prior CAR T therapy or other genetically modified T cell therapy with the exception of subjects who received AMG 119 in this study and are eligible for retreatment.
* Primary immunodeficiency
* History of autoimmune disease resulting in end organ injury or requiring systemic immunosuppression/systemic disease modifying agents within the last 2 years prior to enrollment
* Unresolved toxicities from prior anti-tumor therapy (defined as not having resolved to Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 grade 1, or to levels dictated in the eligibility criteria) with the exception of alopecia or toxicities from prior anti-tumor therapy that are considered irreversible [defined as having been present and stable for > 28 days] which may be allowed if they are not otherwise described in the exclusion criteria AND there is agreement to allow by both the investigator and Amgen
* Received live vaccine within 28 days prior to enrollment
* Exclusion of hepatitis infection based on the following results and/or criteria: Positive for hepatitis B surface antigen (HBsAg) (indicative of chronic hepatitis B or recent acute hepatitis B); Negative HBsAg and positive for hepatitis B core antibody: hepatitis B virus DNA by polymerase chain reaction (PCR) is necessary. Detectable hepatitis B virus DNA suggests occult hepatitis B
* Positive Hepatitis C virus antibody (HCVAb): hepatitis C virus RNA by PCR is necessary. Detectable hepatitis C virus RNA suggests chronic hepatitis C
* History or evidence of any other clinically significant disorder, condition or disease that, in the opinion of the investigator or Amgen physician, if consulted, would pose a risk to subject safety or interfere with the study evaluation, procedures or completion
* Other exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2028-01-14 (Estimated); Study Completion 2028-01-14 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLTs) | Up to 5 years
Incidence of treatment-emergent adverse events and treatment-related adverse events | Up to 5 years
Incidence of clinically significant changes in vital signs | Up to 5 years
Incidence of clinically significant changes in physical examinations | Up to 5 years
Incidence of clinically significant changes in clinical laboratory tests | Up to 5 years

SECONDARY OUTCOMES:
Objective Response (OR) | Up to 5 years
Duration of Response (DOR) | Up to 5 years
Progression-Free Survival (PFS) | Up to 5 years
1-year Overall Survival (1-year OS) | Up to 5 years
Overall Survival (OS) | Up to 5 years
Measurement of expansion and persistence of CAR T cells in peripheral blood post-infusion | Up to 5 years
Evidence of CAR T cells in tumor tissue post dose | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (2):
- United States (2):
  - Research Site, Tampa, Florida
  - Research Site, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Background] Owen DH, Giffin MJ, Bailis JM, Smit MD, Carbone DP, He K. DLL3: an emerging target in small cell lung cancer. J Hematol Oncol. 2019 Jun 18;12(1):61. doi: 10.1186/s13045-019-0745-2. PMID 31215500
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com